CLINICAL TRIAL: NCT06945991
Title: Application and Effect Evaluation of Integrated Nursing and Medical Management in Pediatric Lobar Pneumonia
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Hebei Province (Other)
Responsible Party: Principal Investigator, Linlin Liu, Principal Investigator, Children's Hospital of Hebei Province
Other Study IDs: No. 202222-17
Record Dates: First submitted 2025-04-16; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pediatrics; Lobar Pneumonia; Inflammatory Markers; Satisfaction
MeSH Terms: conditions — Pneumonia; Personal Satisfaction | interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: The control group received routine nursing care
  Interventions: Other: control group
- observation group: the observation group was additionally managed with an integrated nursing and medical approach.
  Interventions: Other: observation group

INTERVENTIONS:
Other: observation group — the observation group was additionally managed with an integrated nursing and medical approach.
  Groups: observation group
Other: control group — The control group received routine nursing care
  Groups: control group

SUMMARY:
Integrated nursing and medical management significantly improves clinical symptoms and pulmonary function in children with lobar pneumonia, shortens hospitalization duration, reduces complication rates, and enhances caregiver satisfaction. These findings support its broad clinical applicability and value.

DETAILED DESCRIPTION:
This study aims to evaluate the clinical efficacy of integrated nursing and medical management in the treatment of pediatric lobar pneumonia. Specifically, it assesses its impact on symptom relief, pulmonary function recovery, inflammatory response control, duration of hospitalization, and caregiver satisfaction. Fifty pediatric patients diagnosed with lobar pneumonia and admitted to our hospital between January and December 2023 were selected and randomly assigned to either the observation group or the control group (n = 25 each) using a random number table. The control group received routine nursing care, while the observation group was additionally managed with an integrated nursing and medical approach. The two groups were compared in terms of duration of fever, cough, pulmonary rales, antibiotic treatment, length of hospital stay, pulmonary function parameters (FEV₁, FVC, FEV₁/FVC), inflammatory markers (CRP, WBC, PCT, LDH), overall treatment efficacy, caregiver satisfaction, and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* (1) Met the diagnostic criteria for lobar pneumonia, presenting with symptoms such as fever, cough, and pulmonary rales, and confirmed by laboratory tests and chest X-ray;
* (2) Aged between 1 and 12 years;
* (3) Informed consent was obtained from the child's legal guardians.

Exclusion Criteria:

* (1)Presence of other concurrent respiratory diseases;
* (2) Congenital or acquired airway malformations, or airway foreign bodies;
* (3) Impaired hepatic or renal function;
* (4) Presence of other systemic diseases;
* (5) Cognitive impairment.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Fifty pediatric patients diagnosed with lobar pneumonia and admitted to our hospital between January and December 2023 were selected and randomly assigned to either the observation group or the control group (n = 25 each) using a random number table.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Time to Clinical Resolution of Symptoms | From admission until discharge (up to 14 days).
  Duration (in days) from hospital admission until resolution of three key symptoms: fever (axillary temperature <37.3°C for 24h), cough (absence of cough for 48h), and pulmonary rales (absence on auscultation). Assessed daily by blinded clinicians.

SECONDARY OUTCOMES:
Change in Pulmonary Function (FEV₁, FVC, FEV₁/FVC) | Baseline (T0) and discharge (T1; up to 14 days).
  Absolute change in spirometry-measured FEV₁ (L), FVC (L), and FEV₁/FVC ratio (%) from admission to discharge. Assessed using standardized spirometry protocols.
Reduction in Inflammatory Markers (CRP, PCT, WBC, LDH) | Baseline (T0) and discharge (T1; up to 14 days).
  Percent reduction in serum CRP (mg/L), PCT (ng/mL), WBC (×10⁹/L), and LDH (U/L) levels from admission to discharge.
Length of Hospital Stay | Up to 14 days.
  Total days from admission to discharge, documented from electronic health records.
Parental Satisfaction Rate | At discharge (T1; up to 14 days).
  Proportion of caregivers reporting "very satisfied" or "satisfied" on a 4-point Likert scale (very satisfied/satisfied/neutral/dissatisfied) at discharge.

OTHER OUTCOMES:
Incidence of Complications | From admission to discharge (up to 14 days).
  Proportion of patients experiencing adverse events (e.g., hemoptysis, pneumothorax, bronchospasm) during hospitalization, verified by imaging/lab reports.
Antibiotic Usage Duration | From admission to discontinuation (up to 14 days).
  Total days of intravenous/oral antibiotic therapy, recorded from medication logs.
Adherence to Rehabilitation Protocols | Daily during hospitalization (up to 14 days).
  Compliance with respiratory exercises (e.g., % of scheduled postural drainage sessions completed), tracked via nursing logs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Children's Hospital, Shijiazhuang, China

REFERENCES:
- [Derived] Hu Y, Guo Q, Liu X, Lv W, Liu L. Integrated nursing and medical management improves outcomes in pediatric lobar pneumonia: a randomized controlled study. Front Pediatr. 2025 Jul 28;13:1612618. doi: 10.3389/fped.2025.1612618. eCollection 2025. PMID 40791810